CLINICAL TRIAL: NCT06975800
Title: Effects of Social Feedback on Intracranial EEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, Tor Wager, Diana L. Taylor Distinguished Professor, Trustees of Dartmouth College
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 467253
Record Dates: First submitted 2025-04-25; First posted 2025-05-16 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Social Influence; Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Patients will watch videos of several doctors. Doctor videos will be presented that increase or decrease expected negative affect (the intervention) in a within-person crossover design.
  Patients will then perform a doctor rating task (reporting on their impressions of warmth, competence, and similar traits associated with care competency).
  Trial blocks consist of a brief video of one of the 8 doctors previously rated by the participant. The doctor will explain what to expect on the upcoming Multimodal Negative Affect Task (MNAT) trials, followed by 4 task trials (fear or math, see Protection of Human Subjects for additional MNAT information). Video cues will include 4 threat-suggestion and 4 safety-suggestion videos for each doctor (8 doctors X 2 low/high threat cues X 3 repetitions x 4 trials per block, 144 total trials).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Random Order 1: Effects of social feedback on intracranial EEG (Experimental): Participants experience trials involving presentation of negative affective stimuli and an effort-demanding cognitive task. Trials are preceded by high or low social cues in random order.
  Interventions: Behavioral: Low social feedback; Behavioral: High social feedback
- Random Order 2: Effects of social feedback on intracranial EEG (Experimental): Participants experience trials involving presentation of negative affective stimuli and an effort-demanding cognitive task. Trials are preceded by high or low social cues in random order.
  Interventions: Behavioral: Low social feedback; Behavioral: High social feedback

INTERVENTIONS:
Behavioral: Low social feedback — Social information is provided to participants signaling that the upcoming trial will be low in negative affect and cognitive effort.
Behavioral: High social feedback — Social information is provided to participants signaling that the upcoming trial will be high in negative affect and cognitive effort.

SUMMARY:
This study aims to assess the impact of social influence on direct neural recordings in human patients undergoing surgical treatment of epilepsy. 24 patients recruited from the Epilepsy Center at Dartmouth Health Medical Center (DHMC) will undergo electrode implantation throughout the brain to localize epileptogenic zones. Patients will be asked to rate their provider's warmth, competence, and other, similar traits associated with care-competency. They will then complete the picture-induced fear and math portions of the multimodal negative affect task (MNAT) during which iEEG is recorded.

DETAILED DESCRIPTION:
This study aims to assess the impact of social influence on direct neural recordings in human patients undergoing surgical treatment of epilepsy. A total of 24 patients, ranging in age from 18 to 65 years, will be recruited from the Epilepsy Center at Dartmouth Health Medical Center (DHMC), which serves a catchment area of approximately 2.5 million people in Northern New England. Patients eligible for intracranial electroencephalography (iEEG) are determined by a clinical-based multidisciplinary board, with 10-20 iEEG studies performed annually in the Epilepsy Monitoring Unit.

Each patient will undergo electrode implantation throughout the brain to localize epileptogenic zones, with 12-20 electrode leads implanted, each containing 8-18 channels. This results in a total of 150 to 220 channels of continuous electrophysiological data per patient. The iEEG signals will be recorded using a Natus clinical system, and precise timing synchronization will be ensured between the iEEG recordings and the experimental paradigm presentation.

The protocol will involve a single one-hour session for each patient. Patients will participate in a doctor rating task, where they provide impressions of warmth, competence, and other qualities related to the doctors presented in the experiment. Additionally, patients will perform a simplified version of the Multimodal Negative Affect Task (MNAT) used in Experiment 2, with the omission of pain stimuli to increase patient acceptability and reduce time and fatigue burden. Trial blocks will consist of brief videos of the doctors explaining what to expect in the upcoming trials, followed by four task trials involving fear or math stimuli from the MNAT task. Each doctor will have four threat-suggestion videos and four safety-suggestion videos, resulting in a total of 144 trials (8 doctors X 2 low/high threat cues X 3 repetitions x 4 trials per block).

The analysis of the neural data will involve time-frequency decomposition of local field potentials (LFPs) to examine broadband gamma-frequency power (40-200 Hz) locked to cue and stimulus onset time. Effects of cues (high vs. low-expectancy), self-reported fear or effort within each cue condition, and their interaction on broadband gamma signals will be assessed for each electrode contact. A focus will be placed on affect-encoding electrodes showing relationships with fear and/or effort within conditions. Proportions of affect-encoding electrodes and other contacts demonstrating social influence effects will be quantified. The analysis will also explore assimilation and contrast effects with cue-predicted values, investigating whether social information influences the neural correlates of affective experience.

To ensure appropriate sample size, it is anticipated that 10-15 eligible patients will participate each year during the project period. Biological sex differences and age will be controlled for in all analyses, and hypotheses will be tested while considering these factors. The study aims to provide valuable insights into the effects of social influence on neural activity, expanding our understanding of the mechanisms underlying placebo effects and affective experiences.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between 18-65 years of age.
* Patients must have a diagnosis of refractory epilepsy undergoing intracranial EEG recording for clinical purposes.
* Patients with a legal guardian will be considered for participation if they are interested and, in the judgment of the research team, they are capable of performing the cognitive tasks required of the study. In those instances, the patient and their legal guardian will both participate in the informed consent process, with the legal guardian signing the consent form.

Exclusion Criteria:

* Patient has additional neurological condition (such as stroke or dementia) or a psychiatric condition (such as active psychosis or suicidal ideation) and are deemed inappropriate for the study.
* Patients are not able to provide informed consent for any reason (e.g. encephalopathic, experiencing a seizure).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Negative affect ratings | Ratings are made 3 to 10 seconds after experiencing each stimulus presented during task performance.
  Participants report subjective negative affect after each trial on a well-validated Generalized Linear Magnitude scale (GLMS) with anchors of "No negative affect" and"Most intense negative affect imaginable". Scale is 0 to 100 with higher values indicating more negative affect.
Cognitive effort ratings | Ratings are made 3 to 10 seconds after experiencing each stimulus presented during task performance.
  Participants report cognitive effort experience after each trial on a well-validated Generalized Linear Magnitude scale (GLMS) with anchors of "No effort" and "Most effort imaginable" . Scale is 0 to 100 with higher values indicating more effort.

SECONDARY OUTCOMES:
Intracranial neural responses to math problems and aversive fear-related images in the amygdala | Continuous recording during task performance, duration 1 hour
  Neural responses will be collected from participants using an iEEG electrode that is implanted by the care team for participant treatment for refractory epilepsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators are strongly committed to contributing to open and reproducible science. All iEEG and behavioral data will be submitted to the NIMH Data Archive (NDA) according to the terms and conditions outlined on their website (https://ndar.nih.gov/contribute_data_sharing_regimen.html ).
  The investigators will ensure that our IRB has approved our Data Sharing Plan. Scientists can use my information, without personal identifiers, for any kind of genetic research.
Time Frame: All data will be de-identified prior to sharing. Raw data will be submitted to NDA within one year from the end of data collection or 6 months from the acceptance date of the first primary study manuscript on the full dataset (excluding methods development papers), whichever is later. Analyzed data/maps of statistical results and models accompanying each paper will be submitted to NDA when the primary study manuscript is accepted.